CLINICAL TRIAL: NCT02062190
Title: Effects of Reveratrol on Cardiovascular Risk Markers and Cognitive Performance in Patients With Schizophrenia: a Randomized Clinical Trilal
Brief Title: Resveratrol, Cardiovascular Risk Markers And Cognitive Performance In Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Karine Zortéa, Master, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RESV-110553; ufrgs110553 (Other: ufrgs)
Record Dates: First submitted 2014-01-15; First posted 2014-02-13 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resveratrol (Active Comparator)
  Interventions: Drug: resveratrol
- corn starch (Placebo Comparator): (10 patients) 100mg 2x/day
  1 month
  Interventions: Drug: resveratrol

INTERVENTIONS:
Drug: resveratrol — 100mg 2x/day
  1 month
  Other Names: Resveratrol (10 patients); Placebo (10 patients)

SUMMARY:
Resveratrol supplementation may improve cardiovascular risk factors and cognitive parameters in patients with schizophrenia taking antipsychotics?

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled trial comparing supplementation with resveratrol or placebo in patients diagnosed with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

Men 18-65 years old, diagnosed with schizophrenia according to DSM-IV and ICD-10, which are in clozapine medication for at least 6 months.

Exclusion Criteria:

Patients will be excluded from the study:

* Have a diagnosis of diabetes
* Use other antipsychotic drugs, clozapine beyond
* Using medicines for diabetes or dyslipidaemia
* Accept not participate in any stage of the research.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Assessment of cardiovascular risk will be realized by measurement of cytokine levels, C-reactive protein and cholesterol levels. | 1 month
  Assessment of cardiovascular risk will be realized by measurement of cytokine levels (IL-12p70, IL-6, IL-10, IL-1b, IL-8 and TNF-α), C-reactive protein and cholesterol levels (total cholesterol, LDL, HDL, triglycerides) in patients with schizophrenia before and after supplementation with resveratrol or placebo.

SECONDARY OUTCOMES:
Cognitive performance will be assessed with a battery of cognitive tests and BPRS (brief psychiatric rating scale) to assess symptoms. | 1 month
  Cognitive performance will be assessed with a battery of cognitive tests (Hopkins, for verbal memory; Stroop: for executive function; Digits WAIS-III, for attention; and Sequence numbers and letters for verbal memory and attention) and BPRS (brief psychiatric rating scale) to assess symptoms.

OTHER OUTCOMES:
Nutritional evaluation will be conducted by anthropometric data and food intake by 24-hour Recall Survey. | 1 month
  Nutritional evaluation will be conducted by anthropometric data (weight, height, waist and hip circumference, body fat percentage) and food intake by 24-hour Recall Survey (24HR).

CONTACTS AND LOCATIONS:
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Zortea K, Franco VC, Francesconi LP, Cereser KM, Lobato MI, Belmonte-de-Abreu PS. Resveratrol Supplementation in Schizophrenia Patients: A Randomized Clinical Trial Evaluating Serum Glucose and Cardiovascular Risk Factors. Nutrients. 2016 Jan 29;8(2):73. doi: 10.3390/nu8020073. PMID 26840331